CLINICAL TRIAL: NCT04876144
Title: You Are Not Alone: a Mobile Application to Reduce Psychosocial Stress
Brief Title: Kogito: App to Reduce Perinatal Psychosocial Stress
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Mental Health, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TL04000197
Record Dates: First submitted 2021-05-02; First posted 2021-05-06 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-04

CONDITIONS: Psychological Stress; Perinatal Problems; Depression, Anxiety
MeSH Terms: conditions — Stress, Psychological; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual care group - clinical (No Intervention): Usual prenatal and postpartum psychiatric care involves regular visits with a psychiatrist from the perinatal psychiatric outpatient clinic of the National Institute of Mental Health, Czechia.
- Usual care group - general (No Intervention): Usual prenatal and postpartum care involves regular visits with one's health care provider while pregnant and after the baby is born.
- Kogito - clinical (Experimental): Usual prenatal and postpartum psychiatric care in perinatal psychiatric outpatient clinic of the National Institute of the National Institute of Mental Health, Czechia plus use of the Kogito app.
  Interventions: Device: Kogito
- Kogito - general (Experimental): Usual prenatal/postpartum care plus use of the Kogito app.
  Interventions: Device: Kogito

INTERVENTIONS:
Device: Kogito — Users of the Kogito app progress throught the deep self-help intervention in a sequence of 5 modules. The base of the Kogito app is in the cognitive-behavioral therapy (CBT), relaxation techniques and peer support.
  Module
  1. Introduction to the CBT (psychoeducation) and deep breathing relaxation plus perinatal peer support videos. Emotional tracking.
  2. Behavioral activization, relaxation techniques, CBT diary, psychoeducation on anxiety and depression, peer support.
  3. CBT - vicious circle, progressive muscle relaxation, peer support content
  4. Cognitive distortions, relaxation in imagination, peer support content
  5. Cognitive restructuring, mindfulness relaxation, peer support content.
  Progress in the Kogito app is conditional on the completion of various CBT tasks
  Arms: Kogito - clinical; Kogito - general

SUMMARY:
The purpose of this research study is to test the efectivness of the remote solution for psychosocial stress in pregnant women and postpartum women. Based on the connection of know-how in the field of social sciences and humanities (psychology, volunteer community and peer work with target group) and technological know-how (software design and development), investigators developed an interactive intervention software (Kogito app) to reduce psychosocial stress in the target group.

DETAILED DESCRIPTION:
This study examine the potential of Kogito app in the delivery of mental and social support care to pregnant and postpartum women using psychometric methods.

A) Clinical efficacy of Kogito app in a clinical cohort. Sample: pregnant or postpartum women with who are being treated in the psychiatric perinatal outpatient clinic of the National Institute of Mental Health, Czech Republic. The app will be tested as a add-on method of care.

Intervention group: Kogito app is added to the usual care Control group: usual care Randomization: 1:1

Participants in the intervention group will be asked to do following things:

1. complete survey questions at entrance into the study
2. use the kogito app
3. complete survey questions one month after study entrance

Participants in the control group will be asked to do following things:

1. complete survey questions at entrance into the study
2. complete survey questions one month after study entrance

B) Clinical efficacy of the Kogito app in a general cohort. The app will be offered free of charge to users from the population of pregnant and postpartum women for the duration of the study.

Recruitment method: advertisements on social networks of National Institute of Mental Health and other public media in Czechia Sample: pregnant or postpartum women from general population in Czechia. The app will be tested using the waiting list as a control condition.

Intervention group: Kogito app Control group: one month waiting list Randomization: 1:1

Participants in the intervention group will be asked to do following things:

1. complete survey questions at entrance into the study
2. use the kogito app
3. complete survey questions one month after study entrance

Participants in the control group will be asked to do following things:

1. complete survey questions at entrance into the study
2. complete survey questions one month after study entrance

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* pregnant women to 1 year after childbirth
* speak, read, and understand Czech
* signing of informed consent to the study and the GDPR form
* participant owns a smart phone and has access to the internet access plus for the clinical group:
* participant is undergoing the usual psychiatric care of the perinatal outpatient clinic of the National Institute of Mental Health, Czechia.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in subjective depression symptoms severity | Baseline to 1 month after study enrollment
  measured by the Edinburgh Perinatal Depression Scale

SECONDARY OUTCOMES:
Change in subjective anxiety symptoms severity | Baseline to 1 month after study enrollment
  measured by the Perinatal Anxiety Screening scale
Change in subjective health related quality of life | Baseline to 1 month after study enrollment
  measured by the Assessment of Quality of Life - eight dimensions scale
Change in subjective loneliness severity | Baseline to 1 month after study enrollment
  measured by the UCLA Loneliness scale 3

CONTACTS AND LOCATIONS:
Overall Officials: Antonin Sebela, MD, PhD, Principal Investigator — National Institute of Mental Health, Klecany, Czechia
Locations (1):
- National Institute of Mental Health, Klecany, Czechia

IPD SHARING:
Plan to Share IPD: No